CLINICAL TRIAL: NCT04165070
Title: KEYMAKER-U01 Substudy 01A: A Phase 1/2, Umbrella Study With Rolling Arms of Investigational Agents With Pembrolizumab With or Without Chemotherapy in Treatment-Naive Participants With Stage IV Non-small Cell Lung Cancer (NSCLC)
Brief Title: KEYMAKER-U01 Substudy 01A: Efficacy and Safety Study of Pembrolizumab (MK-3475) With or Without Chemotherapy When Used With Investigational Agents in Treatment-naïve Participants With Stage IV Non-small Cell Lung Cancer (NSCLC) (MK-3475-01A/KEYMAKER-U01A)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-01A; MK-3475-01A (Other: MSD); KEYMAKER-U01A (Other: MSD); 2023-506932-33-00 (Registry Identifier: EU CT); U1111-1294-6474 (Registry Identifier: UTN); 2020-001626-56 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2019-11-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel; Pemetrexed; patritumab deruxtecan

STUDY DESIGN:
Intervention Model Description: Only participants in Part A will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A: Pembrolizumab+Vibostolimab+Carboplatin + Paclitaxel (Experimental): On Day 1 of each 3-week cycle, participants with squamous NSCLC receive pembrolizumab 200 mg intravenously (IV) PLUS vibostolimab IV PLUS carboplatin Area Under the Concentration-Time Curve (AUC) 6 IV PLUS paclitaxel 200 mg/m^2 IV in Cycles 1-4, followed by maintenance treatment of pembrolizumab 200 mg IV PLUS vibostolimab IV in Cycles 5-35 (total treatment duration: up to approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Biological: Vibostolimab
- Part A: Pembrolizumab+Vibostolimab+Carboplatin + Pemetrexed (Experimental): On Day 1 of each 3-week cycle, participants with nonsquamous NSCLC receive pembrolizumab 200 mg IV PLUS vibostolimab IV PLUS carboplatin AUC 5 IV PLUS pemetrexed 500 mg/m^2 IV in Cycles 1-4, followed by maintenance treatment of pembrolizumab 200 mg IV PLUS vibostolimab IV PLUS pemetrexed 500 mg/m^2 IV in Cycles 5-35 (total treatment duration: up to approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed; Biological: Vibostolimab
- Part A: Pembrolizumab+Boserolimab+Carboplatin+Paclitaxel (Experimental): On Day 1 of each 3-week cycle, participants with squamous NSCLC receive pembrolizumab 200 mg IV PLUS carboplatin AUC 6 IV PLUS paclitaxel 200 mg/m^2 IV PLUS boserolimab IV on Day 1 every 6 weeks (every other 3-week cycle) (Q6W) in Cycles 1-4, followed by maintenance treatment of pembrolizumab 200 mg IV Q3W PLUS boserolimab IV Q6W from Cycles 5 up to Cycle 35 (total treatment duration: up to approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Biological: Boserolimab
- Part A: Pembrolizumab+Boserolimab+Carboplatin+Pemetrexed (Experimental): On Day 1 of each 3-week cycle, participants with nonsquamous NSCLC receive pembrolizumab 200 mg IV PLUS carboplatin AUC 5 IV PLUS pemetrexed 500 mg/m^2 IV PLUS boserolimab IV on Day 1 every 6 weeks (every other 3-week cycle) (Q6W) in Cycles 1-4, followed by maintenance treatment of pembrolizumab 200 mg IV Q3W PLUS pemetrexed 500 mg/m^2 IV Q3W PLUS boserolimab IV Q6W from Cycles 5 up to Cycle 35 (total treatment duration: up to approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed; Biological: Boserolimab
- Part A: Pembrolizumab+MK-4830+Carboplatin+Paclitaxel (Experimental): On Day 1 of each 3-week cycle, participants with squamous NSCLC receive pembrolizumab 200 mg IV PLUS MK-4830 IV PLUS carboplatin AUC 6 IV PLUS paclitaxel 200 mg/m^2 IV in Cycles 1-4, followed by maintenance treatment of pembrolizumab 200 mg IV PLUS MK-4830 IV in Cycles 5-35 (total treatment duration: up to approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Biological: MK-4830
- Part A: Pembrolizumab+MK-4830+Carboplatin+Pemetrexed (Experimental): On Day 1 of each 3-week cycle, participants with nonsquamous NSCLC receive pembrolizumab 200 mg IV PLUS MK-4830 IV PLUS carboplatin AUC 5 IV PLUS pemetrexed 500 mg/m^2 IV in Cycles 1-4, followed by maintenance treatment of pembrolizumab 200 mg IV PLUS MK-4830 IV PLUS pemetrexed 500 mg/m^2 IV in Cycles 5-35 (total treatment duration: up to approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed; Biological: MK-4830
- Part A: Pembrolizumab+MK-0482+Carboplatin+Paclitaxel (Experimental): On Day 1 of each 3-week cycle, participants with squamous NSCLC receive pembrolizumab 200 mg IV PLUS MK-0482 IV PLUS carboplatin AUC 6 IV PLUS paclitaxel 200 mg/m^2 IV in Cycles 1-4, followed by maintenance treatment of pembrolizumab 200 mg IV PLUS MK-0482 IV in Cycles 5-35 (total treatment duration: up to approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Biological: MK-0482
- Part A: Pembrolizumab+MK-0482+Carboplatin+Pemetrexed (Experimental): On Day 1 of each 3-week cycle, participants with nonsquamous NSCLC receive pembrolizumab 200 mg IV PLUS MK-0482 IV PLUS carboplatin AUC 5 IV PLUS pemetrexed 500 mg/m^2 IV in Cycles 1-4, followed by maintenance treatment of pembrolizumab 200 mg IV PLUS MK-0482 IV PLUS pemetrexed 500 mg/m^2 IV in Cycles 5-35 (total treatment duration: up to approximately 2 years).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Biological: MK-0482
- Part B: Pembrolizumab + I-DXd (Experimental): On Day 1 of each 3-week cycle, participants with squamous and nonsquamous NSCLC will receive pembrolizumab 200 mg IV for up to 2 years, PLUS I-DXd in escalating doses until progressive disease or toxicity.
  Interventions: Biological: Pembrolizumab; Biological: Ifinatamab Deruxtecan (I-DXd)
- Part B: Pembrolizumab + Carboplatin + I-DXd (Experimental): On Day 1 of each 3-week cycle, participants will receive pembrolizumab 200 mg IV for up to 2 years, PLUS carboplatin AUC 5-6 up to 4 cycles PLUS I-DXd IV in escalating doses until PD or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Biological: Ifinatamab Deruxtecan (I-DXd)
- Part B: Pembrolizumab + Carboplatin + HER3-DXd (Experimental): On Day 1 of each 3-week cycle, participants will receive pembrolizumab 200 mg IV for up to 2 years, PLUS carboplatin AUC 5-6 up to 4 cycles PLUS HER3-DXd IV in escalating doses until PD or toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Biological: HER3-DXd

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; SCH 900475; KEYTRUDA®
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
  Arms: Part A: Pembrolizumab+Boserolimab+Carboplatin+Paclitaxel; Part A: Pembrolizumab+Boserolimab+Carboplatin+Pemetrexed; Part A: Pembrolizumab+MK-0482+Carboplatin+Paclitaxel; Part A: Pembrolizumab+MK-0482+Carboplatin+Pemetrexed; Part A: Pembrolizumab+MK-4830+Carboplatin+Paclitaxel; Part A: Pembrolizumab+MK-4830+Carboplatin+Pemetrexed; Part A: Pembrolizumab+Vibostolimab+Carboplatin + Paclitaxel; Part A: Pembrolizumab+Vibostolimab+Carboplatin + Pemetrexed; Part B: Pembrolizumab + Carboplatin + HER3-DXd; Part B: Pembrolizumab + Carboplatin + I-DXd
Drug: Paclitaxel — IV infusion
  Other Names: ABRAXANE®
  Arms: Part A: Pembrolizumab+Boserolimab+Carboplatin+Paclitaxel; Part A: Pembrolizumab+MK-4830+Carboplatin+Paclitaxel; Part A: Pembrolizumab+Vibostolimab+Carboplatin + Paclitaxel
Drug: Pemetrexed — IV infusion
  Other Names: ALIMTA®
  Arms: Part A: Pembrolizumab+Boserolimab+Carboplatin+Pemetrexed; Part A: Pembrolizumab+MK-4830+Carboplatin+Pemetrexed; Part A: Pembrolizumab+Vibostolimab+Carboplatin + Pemetrexed
Biological: Vibostolimab — IV infusion
  Other Names: MK-7684
  Arms: Part A: Pembrolizumab+Vibostolimab+Carboplatin + Paclitaxel; Part A: Pembrolizumab+Vibostolimab+Carboplatin + Pemetrexed
Biological: Boserolimab — IV infusion
  Other Names: MK-5890
  Arms: Part A: Pembrolizumab+Boserolimab+Carboplatin+Paclitaxel; Part A: Pembrolizumab+Boserolimab+Carboplatin+Pemetrexed
Biological: MK-4830 — IV infusion
  Arms: Part A: Pembrolizumab+MK-4830+Carboplatin+Paclitaxel; Part A: Pembrolizumab+MK-4830+Carboplatin+Pemetrexed
Biological: MK-0482 — IV Infusion
  Arms: Part A: Pembrolizumab+MK-0482+Carboplatin+Paclitaxel; Part A: Pembrolizumab+MK-0482+Carboplatin+Pemetrexed
Biological: Ifinatamab Deruxtecan (I-DXd) — IV infusion
  Other Names: DS-7300a; MK-2400
  Arms: Part B: Pembrolizumab + Carboplatin + I-DXd; Part B: Pembrolizumab + I-DXd
Biological: HER3-DXd — IV Infusion
  Other Names: U3-1402; MK-1022
  Arms: Part B: Pembrolizumab + Carboplatin + HER3-DXd

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pembrolizumab (MK-3475) with or without chemotherapy in combination with vibostolimab (MK-7684), boserolimab (MK-5890), MK-4830, MK-0482, I-DXd, or HER3-DXd in treatment-naïve participants with advanced squamous or non-squamous NSCLC.

This study is one of the pembrolizumab substudies being conducted under one pembrolizumab umbrella master protocol (MK-3475-U01/KEYMAKER-U01).

DETAILED DESCRIPTION:
The master screening protocol is MK-3475-U01 (KEYMAKER-U01) - NCT04165798

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically- or cytologically-confirmed diagnosis of Stage IV squamous or nonsquamous NSCLC
* Participants with nonsquamous NSCLC who are not eligible for an approved targeted therapy
* Is able to provide archival tumor tissue sample collected either within 5 years or within the interval from completion of last treatment but before entering the screening period or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated obtained within 90 days of treatment initiation
* Has not received prior systemic treatment for their metastatic NSCLC
* Is able to complete all screening procedures within the 35-day screening window for Part A and 28-day screening window for Part B

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a diagnosis of small cell lung cancer
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study treatment administration, or New York Heart Association Class III or IV congestive heart failure
* Has a known history of human immunodeficiency virus (HIV) infection. Well-controlled HIV with anti-retroviral therapy (ART) is not excluded
* Has a known history of Hepatitis B (HPV) or known active Hepatitis C virus infection. Hepatitis B surface antigen (HBsAg) positive is eligible if on HBV antiviral therapy for at least 4 weeks and HBV viral load is undetectable prior to randomization
* Has had major surgery <3 weeks before the first dose of study treatment
* Is expected to require any other form of antineoplastic therapy while on study
* Has a history or current evidence of a gastrointestinal (GI) condition (e.g. inflammatory bowel disease, Crohn's disease, ulcerative colitis) or impaired liver function or diseases that in the opinion of the investigator may significantly alter the absorption or metabolism of oral medications
* Is getting chemotherapy and has clinically active diverticulitis, intra-abdominal abscess, GI obstruction, or peritoneal carcinomatosis
* Has preexisting neuropathy that is moderate in intensity
* Has received prior systemic cytotoxic chemotherapy or other targeted or biological antineoplastic therapy for metastatic disease
* Is unable or unwilling to take folic acid or vitamin B12 supplementation, for participants who will receive pemetrexed
* Has a known sensitivity to any component of carboplatin, paclitaxel, pemetrexed or any of their excipients
* Has received prior radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study treatment
* Has received a live vaccine within 30 days before the first dose of study treatment. Any licensed COVID-19 vaccine (including for Emergency Use) in a particular country is allowed as long as they are messenger ribonucleic acid (mRNA) vaccines, adenoviral vaccines, or inactivated vaccines. Investigational vaccines (ie, those not licensed or approved for Emergency Use) are not allowed
* Has received any prior immunotherapy and was discontinued from that treatment due to a severe or worse immune-related adverse event (irAE)
* Has had chemotherapy or biological cancer therapy within 4 weeks before the first dose of study treatment or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from the AEs due to cancer therapeutics administered more than 4 weeks before the first dose of study treatment (including participants who had previous immunomodulatory therapy with residual irAEs)
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study treatment
* Previously had a severe hypersensitivity reaction to treatment with monoclonal antibodies (including pembrolizumab) and/or any of their excipients
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2032-02-13 (Estimated); Study Completion 2032-02-13 (Estimated)

PRIMARY OUTCOMES:
Part A: Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 24 months
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR will be reported.
Part B: Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 27 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience an AE will be reported.
Part B: Number of Participants Who Discontinue Study Intervention Due to an Adverse Event (AE) | Up to approximately 24 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinue study intervention due to an AE will be reported.
Part B: Number of Participants Who Experience a Dose Limiting Toxicity (DLT) | Up to approximately 3 Weeks
  A DLT is defined as an event with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment that are not due to pre-existing conditions as defined by the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0). Number of participants who experience a DLT per CTCAE 5.0 will be reported.

SECONDARY OUTCOMES:
Part A: Progression-Free Survival (PFS) According to RECIST 1.1 | Up to approximately 24 months
  PFS is defined as the time from first dose of study treatment until either the earliest date of documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS will be reported.
Part A: Number of Participants Who Experience One or More AEs | Up to approximately 27 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience an AE will be reported.
Part A: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 24 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinue study intervention due to an AE will be reported.
Part B: ORR per RECIST 1.1 as assessed by blinded independent central review (BICR) | Up to approximately 24 months
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR will be reported.
Part B: Duration of Response (DOR) per RECIST 1.1 as assessed by BICR | Up to approximately 24 months
  For participants who show confirmed CR or PR, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. DOR will be reported.
Part B: Cmax of I-DXd | At designated time points up to approximately 2 years
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of I-DXd.
Part B: Cmax of HER3-DXd | At designated time points up to approximately 2 years
  Cmax is the maximum concentration of the drug observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of HER3-DXd.
Part B: Cmax of pembrolizumab | At designated time points up to approximately 2 years
  Cmax is the maximum concentration of the drug observed in serum. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax of pembrolizumab.
Part B: Ctrough of I-DXd | At designated time points up to approximately 2 years
  Ctrough is defined as the lowest observed concentration of drug in plasma at the end of the dosing interval. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Ctrough of I-DXd.
Part B: Ctrough of HER3-DXd | At designated time points up to approximately 2 years
  Ctrough is defined as the lowest observed concentration of drug in plasma at the end of the dosing interval. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Ctrough of HER3-DXd.
Part B: Ctrough of pembrolizumab | At designated time points up to approximately 2 years
  Ctrough is defined as the lowest observed concentration of drug in serum at the end of the dosing interval. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Ctrough of pembrolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (46):
- United States (18):
  - Banner MD Anderson Cancer Center ( Site 0001), Gilbert, Arizona
  - City of Hope ( Site 0014), Duarte, California
  - UCSF Medical Center at Mission Bay ( Site 0007), San Francisco, California
  - Georgetown University ( Site 0036), Washington D.C., District of Columbia
  - University of Kentucky Markey Cancer Center ( Site 0019), Lexington, Kentucky
  - MedStar Franklin Square Medical Center ( Site 0033), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 0003), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 0002), Boston, Massachusetts
  - Oncology Hematology West, PC DBA Nebraska Cancer Specialists ( Site 0031), Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center ( Site 0016), Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0037), Hackensack, New Jersey
  - Laura and Isaac Perlmutter Cancer Center ( Site 0034), New York, New York
  - Sanford Fargo Medical Center ( Site 0039), Fargo, North Dakota
  - Cleveland Clinic Main ( Site 0006), Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C ( Site 0015), Columbus, Ohio
  - Abramson Cancer Center of the University of Pennsylvania ( Site 0010), Philadelphia, Pennsylvania
  - Sanford Cancer Center ( Site 0038), Sioux Falls, South Dakota
  - The University of Texas MD Anderson Cancer Center ( Site 0009), Houston, Texas
- Hungary (3):
  - Petz Aladar Megyei Oktato Korhaz ( Site 0062), Győr, Győr-Moson-Sopron
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 0061), Szolnok, Jász-Nagykun-Szolnok
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 0060), Budapest
- Israel (7):
  - Soroka Medical Center ( Site 0072), Beersheba
  - Rambam Health Care Campus-Oncology ( Site 0076), Haifa
  - Shaare Zedek Medical Center ( Site 0075), Jerusalem
  - Meir Medical Center ( Site 0071), Kfar Saba
  - Rabin Medical Center ( Site 0074), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0070), Ramat Gan
  - Sourasky Medical Center ( Site 0077), Tel Aviv
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi ( Site 0173), Florence, Firenze
  - IRCCS Ospedale San Raffaele ( Site 0171), Milan
  - Policlinico Gemelli di Roma ( Site 0174), Roma
- Poland (3):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 0151), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0150), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 0152), Koszalin, West Pomeranian Voivodeship
- South Korea (3):
  - Seoul National University Bundang Hospital ( Site 0081), Seongnam-si, Kyonggi-do
  - Severance Hospital ( Site 0080), Seoul
  - Samsung Medical Center ( Site 0082), Seoul
- Spain (2):
  - ICO L Hospitalet ( Site 0090), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Quiron Madrid ( Site 0091), Madrid
- Taiwan (3):
  - Changhua Christian Hospital ( Site 0181), Changhua
  - Taipei Medical University Hospital ( Site 0180), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0182), Taoyuan District
- Ukraine (4):
  - COMMUNAL NONPROFIT ENTERPRISE "CLINICAL CENTER OF ONCOLOGY, HEMATOLOGY, TRANSPLANTOLOGY AND PALLIATI ( Site 0463), Cherkasy, Cherkasy Oblast
  - Communal Non-Commercial Enterprise "Prykarpatski Clinical On-Surgery department #2 ( Site 0460), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - ME RIVNE REGIONAL ANTITUMOR CENTER ( Site 0461), Rivne, Rivne Oblast
  - Uzhhorod Multispecialty City Clinical Hospital ( Site 0462), Uzhhorod, Zakarpattia Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26292&tenant=MT_MSD_9011